CLINICAL TRIAL: NCT03345446
Title: Circulating RNAs in Acute Heart Failure
Brief Title: Circulating RNAs in Acute Congestive Heart Failure
Acronym: CRUCiAL
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Saumya Das, Co-Director of Resynchronization and Advanced Cardiac Therapeutics Program, Massachusetts General Hospital
Other Study IDs: 2016P001250; 16SFRN29490000 (Other Grant/Funding Number: American Heart Association); 1K23HL127099-01A1 (NIH)
Record Dates: First submitted 2017-08-29; First posted 2017-11-17 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Acute Congestive Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Normal Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood draws collected at the following times and processed for ex-RNAs:
  1. After consent
  2. Prior to discharge
  3. Follow-up within 60 days of leaving the hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with HF-rEF: These patients have Heart Failure with Reduced Ejection Fraction (EF < 55% per the protocol).
  Interventions: Diagnostic Test: Cardiac MRI
- Patients with HF-pEF: These patients have Heart Failure with Preserved Ejection Fraction (EF > 55% per the protocol).
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Cardiac MRI is a test that allows us to look at how the heart muscle works and the amount of scar tissue in your heart. Screening questions will be asked to make sure that patients are not pregnant, and that they have kidney function tests to confirm that IV contrast used (gadolinium) during the MRI is safe for them.

SUMMARY:
The purpose of this American Heart Association-funded and NIH-funded study is to examine circulating RNAs in the acute CHF setting, how they change with decongestive therapy, and their function in vitro and in vivo.

The investigators are testing the hypothesis that ex-RNA levels change significantly during decongestion therapy and can be used as a marker of those individuals who respond to CHF therapy (in terms of cardiac structure or outcome). Additionally, the translational research design allows the investigators to assay the effects of these RNAs on tissue phenotypes in vitro.

DETAILED DESCRIPTION:
Nearly 5 million people in the United States have congestive heart failure (CHF). Although medical therapy such as beta-blockers, angiotensin converting enzyme (ACE) inhibitors, angiotensin-receptor blockers (ARBs) and aldosterone antagonists has improved prognosis, the overall rate of hospital admissions has continued to rise in the last decade and the mortality for patients with symptomatic heart failure remains worse than the majority of cancers in this country. Accordingly, significant opportunities exist for the improvement in outcomes of patients with CHF, both from a morbidity and mortality standpoint. Such opportunities may lie in the outpatient medical management of patients with CHF. Specifically acute CHF represents a particularly underserved area of CHF care.

In this regard, the investigative group and others have demonstrated the utility of extracellular RNAs (short, 20-22 nucleotide RNA molecules stable in circulation in humans) to predict cardiac structural changes and fibrosis in patients post-myocardial infarction with significant changes in cardiac structure. However, little has been done looking at the acute CHF setting. Specific questions include:

1. What RNAs change in the acute CHF setting, and how do these change over time with diuretic therapy?
2. Are these changes in RNA functional? That is, do they cause characteristic changes in the heart in vitro and on heart phenotypes in patients?
3. Do these RNAs predict outcomes in long-term follow-up?

To answer these questions, the investigators will enroll patients who are currently admitted at MGH or BIDMC with acute CHF. The study protocol involves:

1. Venous blood draw, 40 ml anytime within their hospitalization
2. Venous blood draw, 40 ml within 48 hours of planned hospital discharge
3. Venous blood draw, 40 ml at follow-up (within one year of discharge)

Eligible patients (e.g., absence of standard MRI contraindications, GFR > 40ml/min/1.73m2) will be asked pre-discharge or by telephone contact after discharge about coming in for a cardiac MRI study at any point within one year of discharge to examine cardiac structure/function and fibrosis. MRI imaging will be performed by Partners investigators (Dr. Ravi Shah, Dr. Michael Steigner, Dr. Michael Jerosch-Herold) at the 221 Longwood BRIC Imaging Facility (at the Brigham and Women's Hospital, BWH).

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years of age
2. Assessment of LV function within the last year or planned during hospital admission
3. Acute CHF diagnosis, requiring clinical signs and/or symptoms (including exertional or rest dyspnea, orthopnea or PND) AND

   1. N-terminal pro-BNP level > 1000 pg/ml or BNP > 400 pg/ml, OR
   2. Clinical evidence of congestion:

      * X-ray evidence of pulmonary edema or pleural effusions
      * Elevated JVP, lower extremity edema, or rales on pulmonary examination
      * Right heart catheterization evidence of elevated filling pressures (RA pressure > 10 mmHg; PCWP > 18 mmHg)
4. Clinical response to IV diuretic therapy (as judged by a physician)

Exclusion Criteria:

1. Hematocrit at time of consent < 30%
2. End-stage non-cardiovascular diseases

   1. Known HIV/AIDS
   2. Cirrhosis
   3. Hemodialysis-dependent renal failure
3. Pregnancy (as adjudicated by patient history)
4. Ventricular assist device support
5. Acute mechanical support on admission
6. Post-heart transplant
7. Malignancy within the last 1 year or clinically active rheumatologic or autoimmune illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Congestive Heart Failure, either with preserved ejection fraction (HF-pEF) or reduced ejection fraction (HF-rEF).
  The subjects will be enrolled in the acute CHF setting from two sites:
  * Beth Israel Deaconess Medical Center (BIDMC; under direction of Dr. Pablo Pinzon-Quintero, Heart Failure/Transplant Attending Physician)
  * Massachusetts General Hospital (MGH; under direction of Dr. Ravi Shah, Heart Failure/Transplant Attending Physician)
  Subjects will be drawn from the inpatient population at both hospitals, admitted with a diagnosis of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-08-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma RNAs levels (rpm by RNAseq) in patients with acute CHF | admission vs. decongestion (up to 2 weeks)
  Identification of plasma RNAs (absolute reads per million) by RNA sequencing in 1 ml of plasma that are greater than 2 fold increased with p value < 0.05.

SECONDARY OUTCOMES:
Correlation of plasma RNA levels (rpm by RNAseq) with CMR measurements of ventricular function and in vitro fibroblast proliferation assay. | 6 months
  Correlation (by PCA regression models) of candidate plasma RNAs (absolute reads per million) identified in the primary outcome with cardiac MRI phenotypes, including extracellular volume fraction or ECV (unit less), LV ejection fraction (percentage), LV systolic volume (ml) and in vitro fibroblast proliferation by MTT assay (absorbance at 490 nm).

OTHER OUTCOMES:
Correlation of candidate plasma RNA levels (measured by qRT-PCR in fold change compared to endogenous control RNA) with short-term and long-term combined cardiovascular outcome | 4 years
  Correlation of plasma RNA level by sequencing (absolute reads per million) or qRT-PCR (raw CT values, cycle number, or fold change compared to endogenous control, unit-less) with the combined endpoints of mortality, heart failure admissions, or progression to transplantation or LVAD (yes/no) in up to 2-years via review of national death records databases and electronic health care records review.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chatterjee E, Rodosthenous RS, Kujala V, Gokulnath P, Spanos M, Lehmann HI, de Oliveira GP, Shi M, Miller-Fleming TW, Li G, Ghiran IC, Karalis K, Lindenfeld J, Mosley JD, Lau ES, Ho JE, Sheng Q, Shah R, Das S. Circulating extracellular vesicles in human cardiorenal syndrome promote renal injury in a kidney-on-chip system. JCI Insight. 2023 Nov 22;8(22):e165172. doi: 10.1172/jci.insight.165172. PMID 37707956